CLINICAL TRIAL: NCT05595603
Title: Zoledronic Acid-loaded Bone Cement as a Local Adjuvant Therapy for Giant Cell Bone Tumor After Intralesional Curettage: a Prospective, Multicenter, Single Blinded, Randomized Control Trial.
Brief Title: Zoledronic Acid-loaded Bone Cement as a Local Adjuvant Therapy for Giant Cell Bone Tumor After Intralesional Curettage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022_LM1020
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-10

CONDITIONS: Giant Cell Tumor of Bone
Keywords: Zoledronic Acid, intralesional curettage
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — gentamicin-polymethylmethacrylate bead

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zoledronic Acid loaded bone cement (Experimental): 4mg zoledronic acid-loaded gentamicin bone cement (PMMA)
  Interventions: Procedure: 4mg ZOL loaded gentamicin PMMA
- conventional gentamicin bone cement (Active Comparator): gentamicin bone cement (PMMA)
  Interventions: Procedure: gentamicin PMMA

INTERVENTIONS:
Procedure: 4mg ZOL loaded gentamicin PMMA — During surgery, 4mg ZOL will be mixed with gentamicin (1000mg) PMMA cement (40g) by surgeon under sterile conditions to prepare ZOL loaded bone cement, and then it will be filled into the bony defects of the patient where the lesion has been removed after intralesional curettage.
  Arms: Zoledronic Acid loaded bone cement
Procedure: gentamicin PMMA — During surgery, gentamicin (1000mg) PMMA (40g) was prepared by surgeon under sterile conditions and will be filled into the bony defects of the patient where the lesion has been removed after intralesional curettage.
  Arms: conventional gentamicin bone cement

SUMMARY:
The purpose of this study is to investigate whether zoledronic acid-loaded bone cement (4mg ZOL+ gentamicin PMMA ) as adjuvant method can decrease local recurrence in patients with giant cell bone tumor following intralesional curettage surgery. The hypothesis is that patients with local administration of zoledronic acid to the bone cement has lower relapse rate compared those with traditional bone cement(gentamicin PMMA ).

DETAILED DESCRIPTION:
The purpose of the clinical study is to investigate whether the local delivery of zoledronic acid (4mg ZOL-loaded gentamicin PMMA bone cement) as a surgical adjuvant can decrease the local recurrence rate of giant cell tumor (GCT) of bone. The investigators will also evaluate whether patients with zoledronic acid as a surgical adjuvant improves secondary outcomes, including function (MSTS and TESS), surgery related complications (henderson's failure mode) and ZOL-related complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary resectable GCT of bone
* lesion amenable to reconstruction (intralesional curettage) defined as having at least one intact column of bone after removal
* no previous systemic bisphosphonate or denosumab therapy
* with expected longer than 18 months of survival time
* sign the informed consent form

Exclusion Criteria:

* patients with recurrent GCT or extensive GCT which is impossible or inappropriate to use curettage surgery due to its "unresectable" nature.
* conduct unexpected surgery at other center
* the primary goal for surgery is revision
* patient conduct en-bloc/wide resection instead of curettage surgery
* patient can not conduct self-assessment during follow up
* difficulty in complete postoperative follow-up
* previous use of bisphosphonate/ZOL or denosumab drug
* patients have participated in similar research projects
* refused to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
time to first local recurrence | All patients will be followed for this endpoint until 18 months postoperatively
  Time to first local recurrence will be reported during postoperative 18-month follow up period

SECONDARY OUTCOMES:
MSTS score | Doctors will be responsible in filling this questionnaire 3 months, 9 months, 12 months, 18 months postoperatively during patients' follow up
  The Musculoskeletal Tumor Society (MSTS) scoring system is a disease-specific instrument to determine the physical and mental health for patients underwent limb-salvage surgery after tumor resection and is a validated and well-accepted functional scoring system used in orthopaedic oncology research
TESS score | Patients will be asked to fill this survey 3 months, 9 months, 12 months, 18 months postoperatively
  The Toronto Extremity Salvage Score (TESS) is a physical disability measure developed specifically for patients undergoing surgery for extremity tumours and has been shown to have superior measurement properties compared with other commonly used sc
postoperative complication | Patients will be asked to report any complication 1 month, 3 months, 6 months, 9 months, 12 months, 18 months postoperatively during follow up
  Including wound healing problem, mechanical failure, infection and any tumor progression issues
Potential ZOL-related complications | Patients will be followed to report any complication 1 month, 3 months, 6 months, 9 months, 12 months, 18 months postoperatively.
  Patients will be followed for atypical bone fractures and avascular necrosis (AVN) of jaw, one of the most severe complication of ZOL

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No